CLINICAL TRIAL: NCT00985829
Title: Evaluation of Efficacy of Photodynamic Therapy in Basal Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Zohreh Tehranchi-nia, assistant professor of dermatology Shaheed Beheshti Medical University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: pdt bcc1; NCT00985829 (Other Grant/Funding Number: ShaheedBMU)
Record Dates: First submitted 2009-09-26; First posted 2009-09-28 (Estimated); Results first posted 2009-12-22 (Estimated); Last update posted 2009-12-22 (Estimated); Status verified 2009-11

CONDITIONS: Basal Cell Carcinoma
Keywords: basal cell carcinoma; photodynamic therapy; photo chemotherapy; basal cell epithelioma
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Photochemotherapy; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BCC, ALA-PDT (Experimental): Patients with histologically proven basal cell carcinoma who were candidates for treatment with ALA-PDT
  Interventions: Radiation: photodynamic therapy

INTERVENTIONS:
Radiation: photodynamic therapy — treatment of bcc with 5_ALA cream 20% topical administration once monthly+ photodynamic therapy (red light) 120 j/cm2 once monthly
  Other Names: PDT 1200L Waldman Medizintechnik; Schwenningen, Germany

SUMMARY:
The purpose of this study is to evaluate the efficacy of pdt in treatment of bcc and factors that affect response rate.

DETAILED DESCRIPTION:
Background and Aim: Basal cell carcinoma (BCC) is the most common skin cancer .Photodynamic therapy _as a novel , non-invasive therapeutic approach _may be considered a valuable strategy. This study was designed with the aim of the evaluation of efficacy of PDT in treatment of BCC and factors that may affect response rate.

Materials and Methods: This was a clinical trial which was done on 28 BCCs. Patients were treated with ALA-PDT monthly for 1-6 sessions and evaluated for clinical response,cosmetic results and probable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven BCCs

Exclusion Criteria:

* rodent ulcer
* morphea type
* ANA +
* history of photosensitivity or photodermatosis or ingestion of phototoxic drugs during last month
* pregnancy
* breast feeding
* age< 18
* history of another therapeutic intervention for bcc during last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zohreh Tehranchi-nia, assist.prof., Principal Investigator — Skin Research Center

RESULTS

PARTICIPANT FLOW:
Recruitment Details: all patients with Histologically proven basal cell carcinoma (BCC) entered the study.
Pre-assignment Details: Exclusion Criteria:
  rodent ulcer morphea type positive anti nuclear antibody test history of photosensitivity or photodermatosis or ingestion of phototoxic drugs during last month pregnancy breast feeding age< 18 history of another therapeutic intervention for bcc during last 6 months
Groups:
- Aminolevulinic Acid-Photodynamic Therapy (ALA-PDT): Patients with histologically proven basal cell carcinoma who would receive ALA-PDT for their lesion(s)
Period: Overall Study
Arm/Group | Aminolevulinic Acid-Photodynamic Therapy (ALA-PDT)
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Aminolevulinic Acid-Photodynamic Therapy (ALA-PDT)
Number analyzed (Participants) | 28
Age Continuous [Mean (Standard Deviation); unit: years] | 59.1 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response to Photodynamic Therapy
Description: categorized in 3 groups: complete response: there was no visible or palpable lesion; partial response: there was a visible or palpable lesion but the diameter of the lesion had reduced; no response: there was a visible or palpable lesion and the diameter of the lesion had not reduced
Time Frame: immediately after termination of treatment course (with an average of 5 month after initiation of PDT)
Measure: Number; unit: lesions
Groups:
- Aminolevulinic Acid-Photodynamic Therapy (ALA-PDT): Patients with histologically proven basal cell carcinoma who were candidates for photodynamic therapy
Arm/Group | Aminolevulinic Acid-Photodynamic Therapy (ALA-PDT)
Number analyzed (Participants) | 28
lesions
  complete response | 9
  partial response | 14
  no response | 5

2. Secondary Outcome: Histologic Resolution of Lesion
Description: disappearance of the lesion in histologic examination
Time Frame: immediately after the terminaton of treatment course (with an average of 5 months after initiation of PDT)
Population: from those 9 lesions with clinically complete reponse , 3 lesions were biopsied and assessed histologically.
Measure: Number; unit: lesions
Arm/Group | Aminolevulinic Acid-Photodynamic Therapy (ALA-PDT)
Number analyzed (Participants) | 3
lesions
  complete resolution in histologic examination | 3
  not complete resolution in histologic examination | 0

3. Other Pre Specified Outcome: Cosmetic Result
Description: excellent: no scarring, atrophy, or induration, slight or no redness or change in pigmentation compared to the adjacent skin; good: no scarring, atrophy, or induration, moderate redness or increase in pigmentation compared to the adjacent skin; moderate: slight to moderate scarring, atrophy, or induration; and poor: extensive scarring, atrophy, or induration
Time Frame: 1 month after termination of treatment course (with an average of 6 months after initiation of PDT)
Population: cosmetic result was assessed among patients with complete response
Measure: Number; unit: lesions
Arm/Group | Aminolevulinic Acid-Photodynamic Therapy (ALA-PDT)
Number analyzed (Participants) | 9
lesions
  excellent | 5
  good | 2
  moderate | 2
  poor | 0

4. Other Pre Specified Outcome: Location of Lesion
Time Frame: baseline
Measure: Number; unit: lesions
Arm/Group | Aminolevulinic Acid-Photodynamic Therapy (ALA-PDT)
Number analyzed (Participants) | 28
lesions
  scalp | 13
  face | 13
  ear | 2

5. Other Pre Specified Outcome: BCC Type
Description: superficial BCC (sBCC); pigmented BCC(pBCC);nodular BCC (nBCC)
Time Frame: baseline
Measure: Number; unit: lesions
Arm/Group | Aminolevulinic Acid-Photodynamic Therapy (ALA-PDT)
Number analyzed (Participants) | 28
lesions
  nodular | 15
  pigmented | 7
  superficial | 6

6. Other Pre Specified Outcome: Past Medical History of Radiotherapy
Description: past medical history of radiotherapy to the site of tumor before its appearance(for another reason)
Time Frame: baseline
Measure: Number; unit: lesions
Arm/Group | Aminolevulinic Acid-Photodynamic Therapy (ALA-PDT)
Number analyzed (Participants) | 28
lesions
  positive | 17
  negative | 11

ADVERSE EVENTS:
Arm/Group | Aminolevulinic Acid-Photodynamic Therapy (ALA-PDT)
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 2/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aminolevulinic Acid-Photodynamic Therapy (ALA-PDT) (N=28)
local intolerable pain (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes